CLINICAL TRIAL: NCT04513171
Title: A Multi-center, Randomized, Positive-control, Phase 2&3 Combined Study of Y-shape Pegylated Somatropin in Prepubertal Children With Growth Hormone Deficiency.
Brief Title: Safety and Efficacy of Y-shape Pegylated Somatropin in Growth Hormone Deficiency Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Collaborators: Tongji Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TB1805GH
Record Dates: First submitted 2020-08-07; First posted 2020-08-14 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Growth Hormone Deficiency
Keywords: Growth Hormone Deficiency; somatropin; recombinated human growth hormone; Growth Hormone
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Y-shape pegylated somatropin low dose (Experimental)
  Interventions: Drug: Y-shape pegylated somatropin
- Y-shape pegylated somatropin middle dose (Experimental)
  Interventions: Drug: Y-shape pegylated somatropin
- Y-shape pegylated somatropin high dose (Experimental)
  Interventions: Drug: Y-shape pegylated somatropin
- Norditropin-1 (Active Comparator)
  Interventions: Drug: Norditropin®
- Y-shape pegylated somatropin optimal dose (Experimental)
  Interventions: Drug: Y-shape pegylated somatropin
- Norditropin-2 (Active Comparator)
  Interventions: Drug: Norditropin

INTERVENTIONS:
Drug: Y-shape pegylated somatropin — Y-shape pegylated somatropin 100μg/kg, subcutaneous injection, Once weekly.
  Arms: Y-shape pegylated somatropin low dose
Drug: Y-shape pegylated somatropin — Y-shape pegylated somatropin 120μg/kg, subcutaneous injection, Once weekly.
  Arms: Y-shape pegylated somatropin middle dose
Drug: Y-shape pegylated somatropin — Y-shape pegylated somatropin 140μg/kg, subcutaneous injection, Once weekly.
  Arms: Y-shape pegylated somatropin high dose
Drug: Norditropin® — Norditropin 245μg/kg/week, subcutaneous injection, Once daily.
  Arms: Norditropin-1
Drug: Y-shape pegylated somatropin — Y-shape pegylated somatropin 140μg/kg, subcutaneous injection, Once weekly.
  Arms: Y-shape pegylated somatropin optimal dose
Drug: Norditropin — Norditropin 245μg/kg/week, subcutaneous injection, Once daily.
  Arms: Norditropin-2

SUMMARY:
This is a multicenter, randomized, open-labeled, positive controlled phase 2&3 combined study to evaluate the safety and efficacy of weekly Y-shape pegylated somatropin, compared to daily somatropin (Norditropin®), in prepubertal, treatment-naive children with growth hormone deficiency.

DETAILED DESCRIPTION:
This multicenter, randomized, open-labeled, positive controlled study is divided into two stages. The first one is aimed to exploit the optimal dose of Y-shape pegylated somatropin, while the second one is aimed to confirm the efficacy and safety of the study drug. A total of 400 prepubertal children with growth hormone deficiency were expected to enrolled. Subjects will firstly undergo a 52 weeks treatment, and then followed for 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GHD confirmed by two different GH stimulation tests, defined as a peak of GH level of <10.0 ng/ml, determined with a validated assay. Bone age (BA) at least 2 years less than the chronological age. Growth velocity less than 5.0 cm/year. Impaired HT defined as at least 2.0 standard deviations (SD) below of the mean height for chronological age and sex (HT SDS<-2.0).
* Prepubertal (Tanner Ⅰ) males and females by physical examination, aged older than 3 years and younger than10 years for girls and 11 years for boys.
* Short stature with normal intelligence.
* Baseline IGF-1 level below the median IGF-1 level standardized for age and sex.
* Written, signed informed consent of the parent(s) or legal guardian(s) of the subject and written assent of the subject (if the subject is 8 years old or above).

Exclusion Criteria:

* Prior exposure to growth promotion treatment, such as recombinant human growth hormone or gonadal hormones, for more than 1 month.
* Known hypersensitivity to somatropin or excipients, such as mannitol, lysine, sodium chloride.
* Children with closed epiphyses.
* Short stature etiologies other than GHD, such as idiopathic short stature, Turner syndrome, Prader-Willi syndrome, Russell-Silver syndrome, born small for gestational age regardless of GH status.
* Other causes of short stature such as hypothyroidism, adrenocortical hormone deficiency, antidiuretic hormone deficiency.
* Any medical conditions and/or presence that may affect growth velocity such as liver dysfunction, kidney dysfunction, malnutrition, diabetes mellitus, severe dysfunction in major organ such as heart, sever systemic infections, severe immune dysfunction, mental disorders, and other congenital malformations.
* Suffering from chronic infectious diseases such as chronic hepatitis B, AIDS or tuberculosis.
* Receiving non-physiological adrenal corticosteroids.
* Confirmed pituitary and/or hypothalamic malignance by MRI within one year prior to screening. History or presence of any other malignance disease, any evidence of present tumor growth.
* Evidence of congenital intracranial hypertension.
* Evidence of slipped capital femoral epiphysis.
* Evidence of scoliosis over 15°.
* Participation in any other trial of an investigational agent within 3 months prior to screening.
* Any other conditions which in the opinion of the investigator precluded enrollment into the study.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 434 (Actual)
Dates: Start 2018-12-26 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Phase 2: Change of areas under the curve of IGF-1 concentration from baseline (ΔIGF-1 AUC). | 12 weeks
Phase 3: Height velocity. | 52 weeks

SECONDARY OUTCOMES:
Change of height standard deviation score according to chronological age. | 52 weeks
Change of height standard deviation score according to bone age. | 52 weeks
Serum IGF-l level | change from baseline to 52 weeks
Serum IGFBP-3 level | change from baseline to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Luo, MD, Ph.D, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College of HUST, Wuhan, Hubei, China

REFERENCES:
- [Derived] Liang Y, Zhang C, Wei H, Du H, Zhang G, Yang Y, Zhang H, Gong H, Li P, Song F, Xu Z, He R, Zhou W, Zheng H, Sun L, Luo X. The pharmacokinetic and pharmacodynamic properties and short-term outcome of a novel once-weekly PEGylated recombinant human growth hormone for children with growth hormone deficiency. Front Endocrinol (Lausanne). 2022 Aug 11;13:922304. doi: 10.3389/fendo.2022.922304. eCollection 2022. PMID 36034448